CLINICAL TRIAL: NCT03229187
Title: Accurate Prediction and Validation of Response to Neoadjuvant Chemotherapy in Cervical Cancer
Brief Title: Specific Molecular Signatures Predict Neoadjuvant Chemotherapy Response in Cervical Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: Zhejiang University (Other); Wuhan Central Hospital (Other)
Responsible Party: Principal Investigator, Ding Ma, Director of Department of Gynecology and Obstetrics, Huazhong University of Science and Technology
Other Study IDs: 2016-NACT-01
Record Dates: First submitted 2017-07-20; First posted 2017-07-25 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Uterine Cervical Neoplasms; Cervical Cancer; Uterine Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Samples with DNA from blood and tissues.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- neoadjuvant chemotherapy

SUMMARY:
Cervical cancer is one of the major health problems for chinese women. Besides surgery and radiotherapy, neoadjuvant chemotherapy has been proved to be an effective program by many studies.

However, not all patients respond well to neoadjuvant chemotherapy. Knowing the therapeutic effect of the neoadjuvant chemotherapy before receiving it can not only reduce the economic burden, but also more importantly save time to take more suitable treatments.

This study is undertaken to build specific molecular signatures to predict the effects of neoadjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Untreated cervical cancer with FIGO stage Ib-IIb
* Measurable lesions
* Possible to radical hysterectomy
* Age: 18 and older
* Karnofsky Performance Status≥ 70.
* WBC > 3,000/mm³, Hb > 9.0g/dl, Platelet > 100,000 /mm³, SGOT/SGPT < 60 IU/L, T-Bil < 1.5 mg/dL, Cr < 1.2 mg/dL, PaO2 > 80 torr, normal ECG
* Written informed consent

Exclusion Criteria:

* Previous history of cancer
* Patients with previous treatment
* Patients without information of clinical risk factors
* Patients who have active infection

Ages: 18 Years to 70 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patients with histologically confirmed Ib~ IIb cervical carcinoma underwent Neoadjuvant Chemotherapy
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
The clinical response to neoadjuvant chemotherapy | 1 to 3 months
  clinical response（tumor size）

SECONDARY OUTCOMES:
The pathological response to neoadjuvant chemotherapy | 1 to 3 months
  pathological response（<3 mm or not）

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China